CLINICAL TRIAL: NCT00002122
Title: A Randomized Study of Daily and Intermittent Prophylactic Regimens for the Prevention of Disseminated Mycobacterium Avium Complex (MAC) and Fungal Infections in HIV-Infected Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 226A; 066-174
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-04

CONDITIONS: Mycoses; Mycobacterium Avium-Intracellulare Infection; HIV Infections
Keywords: Rifabutin; Mycobacterium avium-intracellulare Infection; Mycoses; Drug Therapy, Combination; Fluconazole; Acquired Immunodeficiency Syndrome; Azithromycin
MeSH Terms: conditions — Mycoses; Mycobacterium avium-intracellulare Infection; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Azithromycin; Rifabutin; Fluconazole

INTERVENTIONS:
Drug: Azithromycin
Drug: Rifabutin
Drug: Fluconazole

SUMMARY:
PRIMARY: To determine the efficacy of azithromycin and rifabutin alone and in combination for the prevention of disseminated Mycobacterium avium Complex (MAC) infection in HIV-infected patients. To determine the efficacy of daily versus weekly fluconazole for the prevention of deep fungal infections in this patient population.

SECONDARY: To determine the incidence of bacterial (including mycobacterial) infections, cryptosporidiosis, and toxoplasmosis in azithromycin versus non-azithromycin containing regimens. To determine the incidence of oropharyngeal and vaginal candidiasis in patients treated with daily versus weekly fluconazole. To compare survival and outcomes of primary endpoints in the treatment arms.

DETAILED DESCRIPTION:
Patients are randomized to receive azithromycin alone, rifabutin alone, or the two drugs in combination for MAC prophylaxis. Patients in each treatment group further receive one of two doses of concomitant fluconazole for deep fungal prophylaxis, unless specifically excluded for fluconazole randomization. Patients are followed for 1 to 2 years.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Preventive therapy with isoniazid for M. tuberculosis.
* Maintenance therapy for CMV retinitis.

Patients must have:

* HIV infection or history of an AIDS-defining condition by CDC criteria.
* One documented CD4 count < 100 cells/mm3 within 12 months prior to study entry.
* NO active MAC disease, MAC bacteremia, or active mycobacterial infection (tuberculous or nontuberculous).
* NO acute opportunistic infection.
* Life expectancy of more than 6 months.
* Consent of parent or guardian if less than legal age of consent.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

ALL PATIENTS -

* Unexplained fevers, elevation in alkaline phosphatase, pancytopenia, abnormal liver function tests, or odynophagia for which the diagnoses of MAC and fungal infections have not been excluded.
* Serious hypersensitivity reactions to macrolides or rifampin.
* Unable to tolerate oral medications. FOR FLUCONAZOLE RANDOMIZATION -
* Serious hypersensitivity reaction to fluconazole.
* Active fungal infection (cryptococcosis, histoplasmosis, blastomycosis, aspergillosis, Candida esophagitis, thrush, vaginal candidiasis).
* Positive baseline urine cryptococcal culture.

Concurrent Medication:

Excluded for fluconazole randomization:

* Maintenance therapy for deep fungal infections.
* Chronic therapy with ketoconazole or fluconazole.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 720

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - UCI Med Ctr, Orange, California
  - UCSD Treatment Ctr / Dept of Medicine and Pediatrics, San Diego, California
  - Santa Clara Valley Med Ctr, San Jose, California
  - Harbor - UCLA Med Ctr, Torrance, California
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - George Washington Univ Med Ctr, Washington D.C., District of Columbia
  - Univ of Massachusetts Med Ctr, Worcester, Massachusetts
  - Univ of Pennsylvania, Philadelphia, Pennsylvania
  - Univ of Texas Southwestern Med Ctr, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Houston Veterans Administration Med Ctr, Houston, Texas

REFERENCES:
- [Background] Havlir DV, Mccutchan JA, Bozzette SA, Dunne M. A double-blind, randomized study of weekly azithromycin, daily rifabutin, and combination azithromycin and rifabutin for the prevention of Mycobactetum avium complex (MAC) in AIDS patients. Conf Retroviruses Opportunistic Infect. 1996 Jan 28-Feb 1;3rd:90